CLINICAL TRIAL: NCT07188688
Title: Shear-Wave Elastography to Detect Enthesitis in Psoriatic Arthritis: Relationship With SIRT2 Expression and Disease Activity
Brief Title: SWE to Detect Enthesitis in PsA: Relationship With SIRT2 Expression and Disease Activity
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Mahmoud Mostafa Nasr Elshenawy, Specialist of Rheumatology, Rehabilitation and Physical Medicine , Assiut University Hospitals, Assiut University
Other Study IDs: SWE of tendons in PsA
Record Dates: First submitted 2025-09-12; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Shear Wave Elastography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Musculoskeletal Ultrasound Device — Musculoskeletal Ultrasound assessment by LOGIQ P10 from General Electric (GE) Healthcare, each patient will be evaluated by grey scale, power doppler MSUS and Shear Wave Elastography (SWE)

SUMMARY:
1. To assess the diagnostic utility of shear-wave elastography (SWE), gray-scale (GS) ultrasound, and Power Doppler (PD) in detecting Patellar and Achilles tendinopathy in psoriatic patients with and without arthritis.
2. Investigate the relation between SWE, GS ultrasound, and PD finding and SIRT2 expression levels.
3. Evaluate the association of the imaging findings and SIRT2 levels with psoriatic arthritis disease activity score.

DETAILED DESCRIPTION:
Psoriatic arthritis is chronic inflammatory arthritis associated with psoriasis which was found in about 20% of patients with psoriatic arthritis. Psoriatic arthritis (PsA) is associated with decreased quality of life. As delayed diagnosis may lead to progressive joint destruction and long-term disability, the key clinical features of PsA should be recognizable to a wide range of clinicians to facilitate early diagnosis. The transition from psoriasis (PsO) to psoriatic arthritis (PsA) and the early diagnosis of PsA is of considerable scientific and clinical interest for the prevention and interception of PsA. Enthesopathy is the cornerstone of the pathophysiology of psoriatic arthritis (PsA). Even in patients without entheses symptoms, enthesitis has been demonstrated by imaging modalities both at the enthesis of load and the so-called "mini-enthesis" (pseudo-enthesis of the fingers). Moreover, inflammatory enthesopathy has been demonstrated in patients with psoriasis (PsO), and it is presumed that this finding could be, to some extent, a predictor of the development of PsA. Psoriatic arthritis is a complex heterogeneous disease manifesting skin disease and several musculoskeletal abnormalities including arthritis, enthesitis, dactylitis and spondylitis. While not all these manifestations are present in every patient, assessment of disease activity should account for these domains. To combining these domains into one composite score has been challenging but several have been developed as Psoriatic Arthritis Disease Activity Score (PASDAS) and Group for Research and Assessment of Psoriasis and Psoriatic Arthritis (GRAPPA) Composite scorE (GRACE index). Musculoskeletal ultrasound (MSUS) imaging plays a pivotal role in the diagnosis and management of musculoskeletal disorders. Additionally, MSUS is a non-invasive, radiation-free and cost-effective tool, making it accessible for routine use in clinical practice. MSUS is playing an increasingly important role in optimizing clinical assessment of patients with rheumatic ultrasound conditions and substantially improves therapeutic and diagnostic capabilities. Ultrasound (US) is a reliable modality in detecting a wide range of musculoskeletal inflammatory lesions in PsA. MSUS correlates well with MRI findings and was found to be more reliable than physical examination in the assessment of musculoskeletal abnormalities. In addition, it is an affordable and accessible tool that is widely used in rheumatology practice. Recent advances in US technology hold promise to introduce highly mobile devices that could potentially be used in non-rheumatology settings (e.g., dermatology, primary care), increasing access to this technology. This highlights the potential use of the US as a point-of-care tool for optimizing early diagnosis of PsA at early stages of their disease. Shear-wave elastography (SWE) is a new technique that provides information on the elastic properties of tissues. It generates the quantitative data in kilopascals (kPa) by measuring the propagation velocity distribution of shear waves in tissues produced by a focused acoustic push pulse. It also provides qualitative data as colour coded images; these images are superimposed on a GS ultrasound image. Harder tissues appear red or yellow and softer tissues appear blue or green. Strain elastography and shear wave elastography reported as shear wave velocity have the best potential to be used in the identification of tendinopathy. Further high-quality studies with robust longitudinal designs to investigate responsiveness are needed to aid the monitoring of tendon recovery. The purpose of the study is to compare the accuracy of SWE with conventional ultrasound (GS and PD) for diagnosing patellar and Achilles tendinopathy in patients with psoriasis with and without arthritis and correlate the findings with clinical symptoms and disease severity scores in patients with psoriasis and psoriatic arthritis. Psoriatic arthritis (PsA) is characterized by a heterogeneous clinical phenotype that makes diagnosis and treatment challenging, particularly in the early stages where diagnosis remains difficult. Currently, diagnosis relies predominantly on clinical findings, highlighting the need for reliable biomarkers to improve diagnostic precision, refine prognostic evaluations, and guide personalized therapeutic strategies. Since a diagnostic delay of more than six months may contribute to poor functional and radiographic outcomes, it is critical to identify biomarkers that can facilitate the early diagnosis of PsA and help predict therapeutic responses. Sirtuins (SIRTs; silent information regulators) are an evolutionarily conserved group of enzymes involved in the post-translational modification of proteins including deacetylation, polyADP-ribosylation, demalonylation and lipoamidation. They exist in many cells and in a variety of organisms. Their names are derived from the SIRT2 (silent information regulator 2) gene, first identified in cells of the yeast Saccharomyces cerevisiae. SIRTs are involved in the recombination of ribosomal DNA and participate in gene silencing and DNA repair. SIRTs are involved in several cellular pathways related to ageing, inflammation, oxidative stress, epigenetics, tumorigenesis, the cell cycle, DNA repair and cell proliferation, positioning them as an essential component in the pathogenesis of many diseases, including psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as PsO by a dermatologist according to PASI score.
* Patients diagnosed as PsA by rheumatologist according to CASPAR classification criteria for psoriatic arthritis
* Adult patients of both sexes with an average > 18 years

Exclusion Criteria:

* Patients with a history of metabolic disease affecting tendons.
* Patients with history of surgery, injury or trauma of patellar and/or Achilles tendon.
* Patients with other rheumatological diseases.
* Patients below 18.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 57 participants: 19 Psoriatic arthritis patients, 19 Psoriasis-only patients and 19 healthy control.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Assessment and comparting the diagnostic utility of shear-wave elastography (SWE) , Gray-scale (GS) ultrasound. and Power Doppler (PD) in detecting tendinopathy in psoriatic patients with and without arthritis. | At baseline (single study visit)
  Musculoskeletal Ultrasound assessment by LOGIQ P10 from General Electric (GE) Healthcare, a division of General Electric Company

SECONDARY OUTCOMES:
Investigate the correlation between SWE, GS ultrasound and PD finding and SIRT2 expression levels and evaluate the correlation of the imaging finding and SIRT2 levels with psoriatic arthritis disease activity score (PASDAS). | At baseline (single study visit)

CONTACTS AND LOCATIONS:
Overall Officials: Eman Abbas M Alkady, Professor, Principal Investigator — Rheumatology, Rehabilitation and Physical Medicine, Assiut University Hospitals; Doaa Kamal M. Abdelhafez, Associate Professor, Principal Investigator — Rheumatology, Rehabilitation and Physical Medicine, Assiut University Hospitals; Nesreen Ismail Ibrahim, Lecturer, Principal Investigator — Rheumatology, Rehabilitation and Physical Medicine, Assiut University Hospitals
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Scalcon MRR, Waclawovsky AJ, Schuch FB, Speeckaert MM, Moresco RN. Proteomic biomarkers in psoriatic arthritis. Clin Chim Acta. 2025 May 15;572:120244. doi: 10.1016/j.cca.2025.120244. Epub 2025 Mar 15. PMID 40096904
- [Background] Saha D, Prakash M, Sinha A, Singh T, Dogra S, Sharma A. Role of Shear-Wave Elastography in Achilles Tendon in Psoriatic Arthritis and Its Correlation with Disease Severity Score, Psoriasis Area and Severity Index. Indian J Radiol Imaging. 2022 Jul 13;32(2):159-165. doi: 10.1055/s-0042-1743116. eCollection 2022 Jun. PMID 35924126
- [Background] Mifsud T, Gatt A, Micallef-Stafrace K, Chockalingam N, Padhiar N. Elastography in the assessment of the Achilles tendon: a systematic review of measurement properties. J Foot Ankle Res. 2023 Apr 27;16(1):23. doi: 10.1186/s13047-023-00623-1. PMID 37101290